CLINICAL TRIAL: NCT04422496
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HEC96719 Tablets in Healthy Subjects
Brief Title: The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of HEC96719 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC96719-P-03
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEC96719 tablets (Experimental): part A: There will be a total of 6 dose cohorts: 0.2 mg, 0.5 mg, 1 mg, 2 mg, 3 mg, and 4 mg part B: There will be a total of 3 dose cohorts: 0.5 mg, 1 mg, 2 mg
  Interventions: Drug: HEC96719
- placebo tablets (Placebo Comparator): part A: There will be a total of 6 dose cohorts: 0.2 mg, 0.5 mg, 1 mg, 2 mg, 3 mg, and 4 mg part B:There will be a total of 3 dose cohorts: 0.5 mg, 1 mg, 2 mg
  Interventions: Drug: HEC96719

INTERVENTIONS:
Drug: HEC96719 — single-Dose Study: Each dose of HEC96719 and placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  multiple-dose study:The study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and multiple-dose study.

SUMMARY:
The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Non-alcoholic fatty liver disease (NAFLD) treatment drug HEC96719 in Healthy Male and Female Subjects

DETAILED DESCRIPTION:
This study consists of a single-dose study and a multiple-dose study, both using a single-center, randomized, double-blind, placebo-controlled, dose-escalation design： I. Single-Dose Study There will be a total of 6 dose cohorts. Each cohort will include 10 subjects, of which 8 receives HEC96719 tablets and 2 receives placebo, regardless of gender. Each subject will only participate in one dose cohort. Each cohort will be divided into 2 group. The first group consists of 2 sentinels, one receiving active and one placebo. The second group will consist of the remainder of the cohort (7 active and 1 placebo) and, following review of the available safety data, will be dosed 48 hours after the sentinel group. Subjects can leave the pharmacy after their biological samples are collected on day 3. The last safety follow-up visit is to be performed on day 7±1 via telephone. Subjects in each cohort will receive a single dose of HEC96719 or placebo in the fasted state on day 1, and safety evaluation is to be performed on day 3 and 7.

II. Multi-Dose Study There will be a total of 3 dose cohorts. Each cohort will consist of 12 subjects, of which 10 receive HEC96719 tablets and 2 receive placebo, the dose regimen will comprise no less than once a day and will not exceed 4 times daily dosing for 7 consecutive days (study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and multiple-dose study). Each subject will only participate in one dose cohort. Subjects will reside at the pharmacy from the day before dosing (D-1) to 96 h after the last dose. Subjects can leave pharmacy after their biological samples are collected. The last safety follow-up visit is to be performed 168±24 h after the last dose via telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 55 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by the Investigator (or designee).
4. Females will be nonpregnant and nonlactating. Females of childbearing potential and male subjects will agree to use contraception
5. Able to comprehend and willing to provide a written Informed Consent Form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. History of gallstone disease or diseases affecting the bile ducts.
5. History of inflammation, ulceration, bleeding affecting the gastrointestinal tract.
6. Alanine transaminase (ALT) or Glutamic oxalacetic transaminase(AST) is out of the normal range.
7. Bilirubin is more than 1.5 x upper limit of normal.
8. Positive test result for hepatitis B surface antigen, hepatitis C virus antibody, and/or human immunodeficiency virus antibodies .
9. History of active tuberculosis or exposure to endemic areas within 8 weeks prior to QuantiFERON®-tuberculosis(TB) testing performed at screening.
10. Positive QuantiFERON®-tuberculosis(TB) indicating possible tuberculosis infection.
11. Immunization with a live attenuated vaccine within 1 month prior to dosing or planned vaccination during the course of the study.
12. History of clinically significant opportunistic infection e.g. invasive candidiasis or pneumocystis pneumonia.
13. Serious local infection e.g. cellulitis, abscess, or systemic infection e.g. septicemia, within 3 months prior to screening.
14. Presence of fever (body temperature >37.6 °C) e.g. a fever associated with a symptomatic viral or bacterial infection, within 2 weeks prior to the first dosing.
15. Subjects who are scheduled to receive an organ transplant or have received an organ transplant;
16. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known), whichever is longer, prior to Check-in.
17. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
18. Use or intend to use any prescription medications/products, within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
19. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
20. History of drug abuse within 1 year prior to screening, or use of soft drugs (such as marijuana) within 3 months prior to the screening, or hard drugs (such as cocaine, phencyclidine, and crack) within 1 year prior to screening.
21. Alcohol consumption of > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL wine), or a positive alcohol breath test at Check-in.
22. Positive urine drugs of abuse screen at Screening or Check-in.
23. Smokers of more than 5 cigarettes per week or positive cotinine test at Screening or Check-in.
24. Consumption of foods and beverages containing poppy seeds, grapefruit, or Seville oranges within 7 days prior to Check-in, consumption of caffeine-containing foods and beverages within 72 hours prior to Check-in, or consumption of alcohol within 48 hours prior to Check-in.
25. Receipt of blood products within 2 months prior to Check-in.
26. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
27. Poor peripheral venous access.
28. Have previously completed or withdrawn from this study, and have previously received the investigational product.
29. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Adverse event | Baseline to day 21
  To assess the safety and tolerability of therapy.

SECONDARY OUTCOMES:
Cmax | predose to 96 hour after dosing
  maximum observed plasma concentration of HEC96719
AUC | predose to 96 hour after dosing
  area under the plasma concentration-time curve (AUC)
T½ | predose to 96 hour after dosing
  apparent terminal elimination half-life
Tmax | predose to 96 hour after dosing
  time of the maximum observed plasma concentration
C4 | predose to 48 hour after dosing
  7α-hydroxy-4-cholestene-3-one
FGF19 | predose to 48 hour after dosing
  Fibroblast growth factor 19
CL/F | predose to 96 hour after dosing
  apparent oral clearance

CONTACTS AND LOCATIONS:
Overall Officials: Jon Rankin, Doctor, Principal Investigator — Study Principal Investigator
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Melbourne VIC 3004, Australia